CLINICAL TRIAL: NCT00407641
Title: Effects of Tinzaparin Sodium on Cardio-vascular OUtcomes and on Blood Lipids in Diabetic Patients on Chronic HEmodialysis: A Long-term, Prospective Study (The "Tinzaparin COULD HELP" Study).
Brief Title: Effects of Tinzaparin on Cardio-vascular Outcomes and on Blood Lipids in Diabetic Patients on Chronic Hemodialysis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Financial and administrative matters did not allow collaboration among centers.
Sponsor: Anemia Working Group Romania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06_06
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-01

CONDITIONS: Diabetes Mellitus; Hemodialysis
Keywords: diabetes mellitus; chronic hemodialysis; anticoagulation; outcome
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Tinzaparin (Experimental): Patients will receive Tinzaparin as anticoagulant during the HD session.
  Interventions: Drug: Tinzaparin administration
- Heparin (Active Comparator): Patients will receive Heparin as an anticoagulant during the HD session
  Interventions: Drug: Heparin administration

INTERVENTIONS:
Drug: Tinzaparin administration — Patients will receive tinzaparin during the HD session
  Arms: Tinzaparin
Drug: Heparin administration — Patients will receive Heparin as an anticoagulant during the HD session.
  Arms: Heparin

SUMMARY:
Low molecular weight heparin (LMWH) provides a safe and effective alternative to UFH for hemodialysis anticoagulation. While unfractionated (UF) heparin has been implicated in hyper-lipidemia, the effect of LMWHs on the lipid profile in non-diabetic patients on chronic hemodialysis remains controversial. The effect of LMWH in diabetic patients, a high risk group for developing hyper-lipidemia and cardio-vascular disease, has not been studied.

The study intends to examine the long-term effects of the replacement of UFH by LMWH (tinzaparin sodium) on cardio-vascular outcomes and on lipoprotein profiles in a large group of diabetic patients stable on HD.

DETAILED DESCRIPTION:
Hemodialysed diabetic patients constitute a high-risk subset of patients for developing cardio-vascular disease, which accounts for nearly 50% of deaths. In those patients, mortality rates probably exceed 20% per year. After stratification for age, race and gender, cardio-vascular mortality is 10-20 times higher in these patients than in the general population. Thus cardio-vascular risk factors in these patients should be managed early, aggressively and in a multi-factorial manner in order to reduce their high cardio-vascular morbidity and mortality.

Low molecular weight heparin (LMWH) provides a safe and effective alternative to UFH for hemodialysis anticoagulation. While unfractionated (UF) heparin has been implicated in hyper-lipidemia, the effect of LMWHs on the lipid profile in non-diabetic patients on chronic hemodialysis remains controversial. The effect of LMWH in diabetic patients, a high risk group for developing hyper-lipidemia and cardio-vascular disease, has not been studied.

The study intends to examine the long-term effects of the replacement of UFH by LMWH (tinzaparin sodium) on cardio-vascular outcomes and on lipoprotein profiles in a large group of diabetic patients stable on HD.

Tinzaparin sodium is superior to UFH in terms of reducing cardio-vascular and cerebrovascular outcomes (primary end-point). Tinzaparin sodium is superior to UFH in terms of reducing the specified lipid parameters of stable diabetic patients on chronic hemodialysis.

A time-to-event analysis is the tool that will be used for recording events rate. Accordingly, the study will aim in enrolling 200 diabetic nephropathy patients, but allowing for a 10% drop-out rate, the number of evaluable patients in the study will be 180.

Therefore, for the primary triple end-point of death/MI/stroke (ischemic) with 180 evaluable patients, we will have an 80% power (at a two-sided alpha level of 0.05) to detect a statistical significant difference in the 2 groups if the rate of events in the UFH group is 30% and on tinzaparin is 13% or less.

For the secondary end-points in cardiovascular morbidity and mortality, if we assume that the event rate in the UFH group is 50%, then a statistical significance can be achieved if the rate in the tinzaparin group is at 30% or less.

For differences in average lipid values between the 2 groups, with 180 evaluable patients, a 2-sided alpha level at 0.05 and with 80% power, we can detect statistical significance if the difference is: for Total Cholesterol=19 mg/dL (SD of 46), for HDL-C = 4.6 mg/dL (SD=11), for TG = 30 mg/dL (SD=72), for LDL-C = 15 (SD=36) and for ApoB = 13 (SD=32).

ELIGIBILITY:
Inclusion Criteria:

* willingness to give written informed consent for participation in the study
* age 18-80 years old
* ability to understand and follow instructions and able to participate in the study for the entire period
* clinically stable (based on the investigator's judgment) within the three months prior to the screening visit
* written and signed agreement

Exclusion Criteria:

* antecedents of cerebrovascular accident, documented myocardial infarction, coronary angioplasty or bypass surgery within 6 months prior to the screening visit
* currently enrollment in any other investigational device or drug study, or participation in another clinical study within 30 days prior to the screening visit
* known or suspected drug or alcohol abuse
* known congenital or acquired bleeding disorders including hepatic failure and amyloidosis, present active major bleeding;
* increased risk of hemorrhage, due to: pericarditis or bacterial endocarditis, severe uncontrolled hypertension, active ulcerative and angiodysplastic gastrointestinal disease, hemorrhagic stroke, shortly after brain, spinal or ophthalmological surgery, concomitant treatment with platelet inhibitors, recent surgical procedures (especially with hemorrhagic complications or those in which hemorrhagic complications would be very severe - cardio-vascular, ophthalmological or neurological), planned surgical procedure within the next week, (history of) heparin-induced thrombocytopenia, with any other disease which, in the opinion of the investigator, makes unacceptable his/her inclusion in the study (known hypersensitivity to heparin, benzyl alcohol, or pork products that should not be treated with innohep®, severe psychiatric disorders, age <18 years, malignant disorders and a life expectancy <6 months, patients that were involved in another research study (studies) in the last month.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
the composite event rate in death (any cause), myocardial infarction and stroke

SECONDARY OUTCOMES:
Cardio-vascular: the composite event rate of unstable angina, transient ischemic attacks, peripheral arterial disease, other, consequent to atherosclerosis
Lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mircescu, Professor, Study Chair — Dr Carol Davila Teaching Hospital of Nephrology; Constantin Verzan, MD, PhD, Study Director — "Dr Carol Davila" Teaching Hospital of Neprology; Cristina Capusa, MD, PhD, Principal Investigator — Dr Carol Davila Teaching Hospital of Nephrology
Locations (13):
- Romania (13):
  - Baia Mare County Hospital, Baia Mare
  - "Sarah" Hemodialysis Centre, Brasov
  - "Dr Carol Davila" Teaching Hospital of Nephrology, Bucharest
  - "N Paulescu" Institute, Bucharest
  - Fundeni Clinical Hospital, Bucharest
  - Cluj University Hospital, Cluj-Napoca
  - Dolj County Hospital, Craiova
  - Vrancea County Hospital, Focşani
  - "CI Parhon" Clinical Hospital, Iași
  - Bihor County Hospital, Oradea
  - Prahova County Hospital, Ploieşti
  - Dambovita County Hospital, Târgovişte
  - Timisoara County Hospital, Timișoara

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593